CLINICAL TRIAL: NCT05890742
Title: A Phase 1b/3 Clinical Trial Evaluating the Efficacy and Safety of IBI310 in Combination With Sintilimab, for Neoadjuvant Treatment of Microsatellite Instability-high or Mismatch Repair-deficient, Resectable Colon Cancer
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of IBI310 in Combination With Sintilimab, for Neoadjuvant Treatment of MSI-H/dMMR Resectable Colon Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310L301
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: MSI-H
Keywords: dMMR; resectable colon cancer
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase Ib Experimental group (Experimental): In Phase Ib Experimental group，subjects will receive two cycles of neoadjuvant immunotherapy: the first cycle of IBI310 (1mg/kg) & Sintilimab (200mg) and the second cycle of Sintilimab (200mg) only.Followed by radical surgery for colon cancer.
  Interventions: Drug: IBI310&Sintilimab; Procedure: Radical surgery
- Phase Ib Control group (Active Comparator): In Phase Ib Control group，subjects will receive two cycles of neoadjuvant immunotherapy with 200 mg of sintilimab per cycle, followed by radical surgery for colon cancer.
  Interventions: Drug: Sintilimab; Procedure: Radical surgery
- Phase III Experimental group (Experimental): In Phase III Experimental group，subjects will receive two cycles of neoadjuvant immunotherapy: the first cycle of IBI310 (1mg/kg) & Sintilimab (200mg) and the second cycle of Sintilimab (200mg) only. Followed by radical surgery for colon cancer. Adjuvant chemotherapy will be given or not according to the pathological stage after surgery.
  Interventions: Drug: IBI310&Sintilimab
- Phase III Control group (Active Comparator): In Phase III Control group, subjects will receive radical surgery without neoadjuvant therapy. Adjuvant chemotherapy will be given or not according to the pathological stage after surgery.
  Interventions: Procedure: Radical surgery

INTERVENTIONS:
Drug: Sintilimab — In ARM Phase Ib Control group, Sintilimab will be used twice, q3w.
  Arms: Phase Ib Control group
Drug: IBI310&Sintilimab — In ARM Phase Ib&III Experimental group，IBI310&Sintilimab will be used in first cycle, Sintilimab will be used in second cycle(q3w). Radical surgery after neoadjuvant therapy.
  Arms: Phase III Experimental group; Phase Ib Experimental group
Procedure: Radical surgery — In ARM Phase Ib&III Experimental group, Phase Ib Control group, subjects will receive radical surgery after neoadjuvant therapy. In ARM Phase III Control group,subjects will receive radical surgery without neoadjuvant therapy
  Arms: Phase III Control group; Phase Ib Control group; Phase Ib Experimental group

SUMMARY:
Evaluate efficacy and safety of IBI310 (CTLA-4 antibody) in combination with Sintilimab, for neoadjuvant treatment of MSI-H/dMMR resectable colon cancer

ELIGIBILITY:
Inclusion Criteria:

1. Signed the Informed Consent Form (ICF) and complied with the visit and related procedures stipulated by the plan;
2. At least 18 years old.
3. Primary colon adenocarcinoma was histologically confirmed.
4. Radiographic assessment showed a resectable stage IIB-III based on AJCC Stage VIII (cT4 or cN+ only).
5. MSI-H or dMMR.
6. Radical excision can be performed before neoadjuvant therapy after diagnosis by the investigator.
7. Have at least one evaluable lesion according to the RECIST v1.1 evaluation criteria.
8. The Eastern Cooperative Oncology Group performance status (ECOG PS) is 0 to 1.

Exclusion Criteria:

1. Previously received any antitumor therapy for the disease under study, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.
2. Prior treatment with anti-PD-1, anti-PD-L1, anti-programmed death receptor ligand 2 (PD-L2) or anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) or any other drug acting on T-cell co-stimulation or immune checkpoint pathways (such as OX40, CD137, etc.) and adoptive cellular immunotherapy.
3. Concurrent participation in another clinical study, unless participating in an observational (non-interventional) clinical study or in the survival follow-up phase of an interventional study.
4. Received any investigational drug or device treatment within 4 weeks prior to initial administration of the investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2028-04-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response(pCR), defined as the proportion of subjects with no residual tumor in the primary tumor removed and in all lymph nodes removed after neoadjuvant therapy. | 1 month after surgery
  The proportion of subjects with no residual tumor in the primary tumor removed and in all lymph nodes removed after neoadjuvant therapy.
Event Free Survival, EFS(EFS), defined as the time from randomization to the first determination using RECIST v1.1 of inoperable disease progression, local recurrence or distant metastasis after surgery, or death from any cause, whichever occurs first. | up to 5 years after surgery
  The time from randomization to the first determination using RECIST v1.1 of inoperable disease progression, local recurrence or distant metastasis after surgery, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
R0 tumor resection rate, defined as the proportion of subjects with R0 excision | 2 week after surgery
  The proportion of subjects with R0 excision
Overall-survival(OS), defined as the time from randomization to death from any cause | up to 5 years after surgery
  The time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China